CLINICAL TRIAL: NCT06849830
Title: Incorporating Narrative Into the Treatment of Youth With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-43017
Record Dates: First submitted 2025-02-08; First posted 2025-02-27 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative Medicine (NM) Workshop Series (Experimental): Participants in this study will take part in a six-week Narrative Medicine (NM) curriculum designed to enhance self-expression, reflection, and resilience in individuals with anorexia nervosa. Workshops will be conducted weekly at the UCSF Eating Disorders Program and will include:
  * Close reading of visual or written texts related to themes such as self-definition, resilience, kindness, and possibility
  * Creative writing exercises in response to structured prompts
  * Group discussions and sharing to foster community, connection, and self-expression
  Interventions: Behavioral: Narrative Medicine (NM) Workshop Series

INTERVENTIONS:
Behavioral: Narrative Medicine (NM) Workshop Series — The Narrative Medicine (NM) Workshop Series is a structured six-week behavioral intervention designed to enhance self-expression, reflection, and resilience in adolescents and young adults recovering from eating disorders. This intervention differs from traditional psychotherapeutic or psychoeducational approaches by integrating literary analysis, creative writing, and guided discussion as therapeutic tools.
  Each one-hour weekly workshop includes:
  * Close reading of visual or written texts related to themes such as self-definition, resilience, kindness, and possibility
  * Creative writing exercises in response to structured prompts that encourage self-reflection and personal storytelling
  * Facilitated group discussions to foster connection, self-expression, and emotional processing in a supportive environment

SUMMARY:
The goal of this clinical trial is to evaluate whether a narrative medicine (NM) curriculum can enhance self-expression, reflection, and resilience in adolescents and young adults with anorexia nervosa.

The main questions it aims to answer are:

* Does participation in an NM curriculum improve self-expression and reflection in individuals with anorexia nervosa?
* Does engaging in creative writing and group discussion promote resilience and emotional processing in this population?

Participants will be 16-25 years old, medically stable for outpatient eating disorder therapy, and actively engaged in treatment. Those with active suicidal ideation, recent non-suicidal self-injury, or a co-occurring personality disorder will not be eligible.

Participants will:

* Attend six weekly workshops (April-May 2025) focused on themes such as self-definition, kindness, resilience, and possibility
* Engage in close reading of visual or written texts
* Complete creative writing exercises in response to prompts
* Participate in group discussions and sharing

An optional capstone reading event will provide a supportive space for participants to share their work with peers, loved ones, and providers, fostering connection and community.

This study aims to explore the role of narrative medicine in eating disorder treatment and assess its potential benefits for psychological well-being and self-expression.

ELIGIBILITY:
Inclusion Criteria:

* 16-25 years old
* have a DSM-5 diagnosis of AN (confirmed by the UCSF Eating Disorders Program clinical team),
* currently engaged in outpatient eating disorder treatment, ensuring medical stability and capacity for a group-based intervention
* English fluency to engage in reflective writing and discussions
* Cognitive ability to meaningfully participate in narrative-based exercises

Exclusion Criteria:

* Currently medically unstable or require inpatient hospitalization
* History of psychosis, schizophrenia spectrum disorder, bipolar disorder, or personality disorder
* Severe neurocognitive impairment that would prevent engagement with the intervention
* Active suicidal ideation or non-suicidal self-injury within the past two months
* Insufficient English proficiency to participate in group discussions and writing exercises

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants in each session | Immediately post-intervention (Week 6)
  Feasibility will be measured by participant retention in intervention.
Satisfaction with intervention components using 5-point Likert scales and semi-structured individual interviews | Immediately post-intervention (Week 6)
  Acceptability will be measured by questionnaire including 5-point Likert scales and semi-structured individual interviews assessing content relevance, writing prompts, group discussions, and facilitation.
  Scale title: Intervention Satisfaction Questionnaire (ISQ) Minimum value: 1 (Strongly Disagree) Maximum value: 5 (Strongly Agree) Interpretation: Higher scores indicate greater satisfaction with the intervention (better outcome).

SECONDARY OUTCOMES:
Identity Clarity | Pre- (Week 0) and immediately post-intervention (Week 6)
  Assessed using the Erikson Psychosocial Stage Inventory - Identity Subscale (EPS-Identity), which evaluates self-concept clarity and personal identity coherence.
  Scale title: Erikson Psychosocial Stage Inventory - Identity Subscale (EPS-Identity) Minimum value: 1 (Strongly Disagree) Maximum value: 5 (Strongly Agree) Interpretation: Higher scores indicate stronger identity development and consolidation (better outcome).
Social Connectedness | Pre- (Week 0) and immediately post-intervention (Week 6)
  Measured using the Social Connectedness Scale (SCS), which assesses perceived closeness to others and sense of belonging.
  Scale title: Social Connectedness Scale (SCS) Minimum value: 1 (Strongly Disagree) Maximum value: 6 (Strongly Agree) Interpretation: Higher scores indicate greater feelings of social connectedness and belonging (better outcome).
Depression Symptoms | Pre- (Week 0) and immediately post-intervention (Week 6)
  Measured using the Patient Health Questionnaire-9 (PHQ-9) for depressive symptoms.
  Scale title: Patient Health Questionnaire-9 (PHQ-9) Minimum value: 0 (Not at all) Maximum value: 3 (Nearly every day) Interpretation: Higher scores indicate greater severity of depressive symptoms (worse outcome).
Anxiety Symptoms | Pre- (Week 0) and immediately post-intervention (Week 6)
  Measured using the Generalized Anxiety Disorder-7 (GAD-7) for anxiety.
  Scale title: Generalized Anxiety Disorder 7-item (GAD-7) Scale Minimum value: 0 (Not at all) Maximum value: 3 (Nearly every day) Interpretation: Higher scores indicate greater severity of anxiety symptoms (worse outcome).
Eating Disorder Severity | Pre- (Week 0) and immediately post-intervention (Week 6)
  Measured using the Eating Disorder Examination Questionnaire (EDE-Q), which captures cognitive and behavioral symptoms of AN, and percent of expected body weight (EBW) at follow-up.
  Scale title: Eating Disorder Examination Questionnaire (EDE-Q) Minimum value: 0 (No days / Not at all) Maximum value: 6 (Every day / Extremely) Interpretation: Higher scores indicate greater severity of eating disorder psychopathology (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Anoushka Sinha, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Nancy Friend Pritzker Psychiatry Building, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knio L, Sridhar H. Phenomenology of Identity: Narrative Medicine Curricula in the Care of Eating Disorders. J Med Humanit. 2025 Dec;46(4):673-696. doi: 10.1007/s10912-025-09929-6. Epub 2025 Jan 27. PMID 39869237